CLINICAL TRIAL: NCT05536050
Title: Prospective Observational Pilot Study of Low-dose Naltrexone in Patients With Chronic Migraine With Comorbid Fibromyalgia
Brief Title: Study of Low-dose Naltrexone in Chronic Migraine With Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 22D.486
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Chronic Migraine; Fibromyalgia; New Daily Persistent Headache
MeSH Terms: conditions — Fibromyalgia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Migraine diary and Questionnaires — Patients who already have a prescription for low-dose naltrexone will be administered questionnaires twice during the trial. Additionally, patients will maintain migraine diary for the duration of the trial.

SUMMARY:
This research aims to look at the effect of low-dose naltrexone on the severity and frequency of attacks in people with chronic migraine with or without new daily persistent headache and fibromyalgia. A few studies suggest low-dose naltrexone is effective for fibromyalgia, but it has not been studied in patients with migraine and headaches. Our goal is to see if there is an improvement in either severity and frequency of attacks and overall impact on quality of life over a three-month period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be adults of all genders ages 18 and older.
* Patients with a diagnosis of CM (with or without NDPH) by IHC-3 criteria, diagnosed by a certified headache specialist.
* Subjects who received a new prescription for LDN
* Fibromyalgia-diagnosed according to Fibromyalgia Rapid Screening Tool
* Subjects should be on stable headache and migraine preventives for the past 2 months with no plans to change medication for the next 4 months.
* Subjects willing to maintain a headache/migraine diary one month prior to taking medication and while taking the medication, either physical or electronic diary of their choice.
* Subjects willing to fill out pre and post intervention surveys
* Subjects willing to comply with planned follow up phone calls and visits.

Exclusion Criteria:

* Not planning on follow up care with clinician.
* Patients with decreased decision-making capacity in which the investigator's opinion would interfere with the person's ability to provide informed consent and complete study questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be screened and enrolled by study personnel either during their visit with their referring physician, or remotely.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness on migraine | 9-12 weeks
  Monthly migraine days

SECONDARY OUTCOMES:
Effectiveness on headache | 9-12 weeks
  Monthly headache days
Intensity | 9-12 weeks
  Average peak intensity of migraine
The Migraine Disability Assessment Test | 9-12 weeks
  Impact of migraine on daily life
Migraine Specific Quality of Life Index | 9-12 weeks
  Impact of migraine and migraine treatment on quality of life
Patient Health Questionnaire | 9-12 weeks
  Monitor depression and changes in signs/symptoms of depression
Fibromyalgia Impact Questionnaire | 9-12 weeks
  Assess health status of patients with fibromyalgia
Patients' Global Impression of Change | 9-12 weeks
  Assess patient's belief in efficacy of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No